CLINICAL TRIAL: NCT05721677
Title: The Impact of Central-line Exit-site Sealing With 2-octyl Cyanoacrylate Adhesive on CLABSI in Pediatric Cardiac Intensive Care Unit
Brief Title: CLABSI Prevention With Tissue Adhesive
Acronym: Cya-No-CLABSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, ERAN SHOSTAK, Principal Investigator, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RMC220375CTIL
Record Dates: First submitted 2023-01-17; First posted 2023-02-10 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Central-line Associated Blood Stream Infections (CLABSI)
Keywords: CLABSI; Pediatric; Cardiac intensive care; cyanoacrylate; tissue adhesive

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open labeled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tissue adhesive (Experimental): Tissue adhesive application at the CVL exit-site, on all CVLs, PICCs during the patient LOS. Regular CLABSI preventive protocol. Regular preventive CVL dressings (Chlorhexidine >2mo).
  Interventions: Device: 2-octyl cyanoacrylate based topical skin adhesive
- Control group (No Intervention): Regular CLABSI preventive protocol. Regular preventive CVL dressings (Chlorhexidine >2mo).

INTERVENTIONS:
Device: 2-octyl cyanoacrylate based topical skin adhesive — Tissue adhesive on CVL exit-site
  Arms: Tissue adhesive

SUMMARY:
Our aim is to test the effect of tissue adhesive application at the Central-line exit-site on CLABSI rates in high-risk pediatric congenital heart disease patients.

DETAILED DESCRIPTION:
Health-care associated infections (HAI) and especially central-line associated blood stream infections (CLABSI) are a well described burden in the intensive care units. There are two main possible pathways leading to central-venous line (CVL) related infection: the first is migration of microbes down the catheter tract (between the CVL and the skin), and the second is via the catheter hub/lumen. Cyanoacrylate adhesive is a commonly used tissue adhesive in children and adults with frequent use in pediatric facial lacerations. Several studies have shown its feasibility and safety in the general pediatric population, including neonates and in children after cardiac surgery.

To our knowledge, no study to date has explored the use of 2-octyl cyanoacrylate at central-line exit site as a mean to decreases pediatric CLABSI.

Our aim is to assess 2-octyl cyanoacrylate association with CLABSI rate in pediatric cardiac intensive care population.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to pediatric cardiac ICU (PCICU) defined as high-risk for CLABSI (any of):

* young age<1y & Congenital Heart Surgery Mortality Category (STAT\STS-EACTS) score 2-5
* Risk Adjustment for Congenital Heart Surgery (RACHS) category ≥3
* preoperative length-of-stay (LOS) >7 days
* preoperative ventilator support
* presence of a genetic abnormality
* extracorporeal membrane oxygenation (ECMO) support

Exclusion Criteria:

* Patients with on-going bacteremia
* patients with pre-existing central-line or peripherally inserted central catheter (PICC)
* parental refusal to participate.

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
CLABSI rate | up to 1 year

SECONDARY OUTCOMES:
dressing changes rates | average of 14 days
safety outcome: Number pf participants with contact dermatitis at the catheter exit site, line dislodgement, leak, exit site bleeding, allergic reaction or line tunnel infection | average of 14 days
  number of patients suffering from contact dermatitis at the catheter exit site, line dislodgement, leak, exit site bleeding, allergic reaction or line tunnel infection
invasive mechanical ventilation duration | up to 1 year
  days
ICU LOS | up to 1 year
  days
Postoperative ECMO support | up to 1 year
Chylothorax | up to 1 year
Chest drains duration | up to 1 year
  days
need for cardiopulmonary resuscitation (CPR) | up to 1 year
Extubation failure | up to 1 year
  rate
presence of lung atelectasis | up to 1 year
multidrug resistant bacterial colonization | up to 1 year
mortality rate | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ovadia Dagan, Prof. M.D, Study Director — Director PCICU, Schneider Children's Medical Center
Locations (1):
- Schneider's children medical center, Petah Tikva, Israel